CLINICAL TRIAL: NCT06412341
Title: A Feasibility Study to Inform an RCT to Evaluate 'Accepting Your Body After Cancer', an Online-delivered, Group-based CBT Body Image Intervention, for Women Who Have Received Treatment for Breast Cancer
Brief Title: Feasibility Study of ABC for Women Treated for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10473704
Record Dates: First submitted 2024-04-25; First posted 2024-05-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Female
Keywords: Body Image; Feasibility; Intervention; Cognitive Behavioural Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABC + Macmillan body image booklet (Experimental): Accepting your Body after Cancer (ABC) + Macmillan Cancer Support psycho-educational body image booklet
  ABC comprises seven 2-hour group sessions (with approximately 8 women per group) delivered online via Microsoft Teams and across 7 consecutive weeks. The intervention aims to improve body image among women treated for BC. Rooted in CBT, ABC uses strategies to alter unhelpful thoughts, reduce anxiety, and promote non-avoidant behaviours. Other topics are also explored, including sociocultural pressures for women, intimacy, physical activity, self-care, mindfulness, and relaxation. The sessions will be guided using PowerPoint slides, which will include text, images, and videos. Each session will include individual and group-based activities, and participants will be asked to complete between-session readings and activities. (Macmillan Cancer Support psycho-educational body image booklet is described below).
  Interventions: Behavioral: Accepting your Body after Cancer; Behavioral: Macmillan body image booklet
- Macmillan body image booklet (usual care) (Other): Macmillan Cancer Support psycho-educational body image booklet (only)
  Discussions with PPI advisors indicated that some form of body image-specific support should be provided for the control arm. Macmillan's freely available psychoeducational body image booklet was considered appropriate, given that the thorough 77-page booklet provides a substantial amount of support and guidance relating to managing body image concerns. It explains the effects of cancer on body image, and provides practical guidance (e.g., make-up) and psychoeducational guidance (e.g., managing others' reactions), in addition to some CBT strategies. Upon randomisation to the control arm, participants will be sent the Macmillan body image booklet and encouraged to work through it gradually. The booklet can be accessed via the following webpage: https://cdn.macmillan.org.uk/dfsmedia/1a6f23537f7f4519bb0cf14c45b2a629/791-source/body-image-mac14192
  Interventions: Behavioral: Macmillan body image booklet

INTERVENTIONS:
Behavioral: Accepting your Body after Cancer — See 'Arm Description'
  Arms: ABC + Macmillan body image booklet
Behavioral: Macmillan body image booklet — See 'Arm Description'

SUMMARY:
The investigators aim to assess the feasibility and acceptability of conducting a randomised controlled trial (RCT) to test whether receiving ABC (an online-delivered, Cognitive Behavioural Therapy [CBT], group-based, body image programme) alongside a psychoeducational body image booklet provides greater benefits to women treated for breast cancer compared to a receiving a psychoeducational body image booklet alone.

Results from this feasibility study will inform the design, management, and future delivery of a definitive randomised controlled trial to assess effectiveness and cost-effectiveness of ABC.

Specific objectives are to:

* Establish appropriate, inclusive, and acceptable methods of participant recruitment, retention, and management procedures.
* Establish the feasibility and acceptability of quantitative data collection, including determining appropriate primary and secondary outcome measures.
* Adapt and test a measure of health and social care service use, to inform a future economic evaluation.
* Establish intervention adherence and acceptability (of online setting) among participants and ABC facilitators.

Participants will be randomised to either the intervention or control arm. The control arm will receive the Macmillan Cancer Support psychoeducational body image booklet. The intervention arm will receive the Macmillan booklet and the ABC programme, a 7-session, CBT group-based programme delivered online. All participants will complete self-report validated outcome measures at weeks 1 (T1; baseline/pre-intervention), 9 (T2; immediate post-intervention), 20 (T3; three-month post intervention), and 32 (T4; six-month post intervention). Following drop-out or completion of all study procedures, a subset of participants will be invited to take part in interviews.

DETAILED DESCRIPTION:
BACKGROUND

Breast cancer is the most common cancer among women in the UK, with 55,500 diagnosed annually. Fortunately, 85% live at least five years following their diagnosis, however, they live with treatment-related consequences, including changes to the body, such as breast asymmetry, hair loss/thinning, and fatigue. These changes adversely impact body image.

Body image distress among this group is pervasive, with little improvement five years post-treatment. Further, its consequences of anxiety, depression, sexual/intimacy issues, poorer quality of life, and shorter survival, warrant attention, as these psychosocial concerns are higher among UK-based breast cancer survivors versus women with no cancer history. This is costly for society, as depression and anxiety among women treated for breast cancer lead to greater healthcare use and costs, and economic losses.

The above emphasises the need to target body image distress among women treated for breast cancer. However, the investigators conducted a systematic review of body image interventions for this group, which revealed a gap regarding interventions with lasting improvements. This highlighted the need to develop an effective body image intervention for this group, and thus informed the development of our intervention, 'Accepting your Body after Cancer' (ABC).

Preliminary data indicates that ABC shows promise. However, online delivery of ABC may overcome barriers, increase geographic accessibility and, and thus, facilitate inclusion of women from diverse backgrounds and reduce health inequalities. Such online delivery would also be less costly than in person delivery and will facilitate sustainability of the intervention. Prior to a full-scale RCT to establish the effectiveness of online ABC delivery, a feasibility study is needed to ensure appropriate study design parameters.

AIMS AND OBJECTIVES

The investigators aim to assess the feasibility and acceptability of conducting an RCT to test whether receiving ABC alongside a psychoeducational body image booklet provides greater benefits to women treated for breast cancer compared to a receiving a psychoeducational body image booklet alone.

Results from this feasibility study will inform the design, management, and future delivery of a definitive randomised controlled trial to assess effectiveness and cost-effectiveness of ABC.

Specific objectives are to:

* Establish appropriate, inclusive, and acceptable methods of participant recruitment, retention, and management procedures.
* Establish the feasibility and acceptability of quantitative data collection, including determining appropriate primary and secondary outcome measures.
* Adapt and test a measure of health and social care service use, to inform a future economic evaluation.
* Establish intervention adherence and acceptability (of online setting) among participants and ABC facilitators.

This study will examine uncertainties that need addressing before a definitive RCT:

* Recruitment processes and response rates: Responses from potential participants invited for randomisation and investigating reasons for declining.
* Intervention adherence and retention within the study: Percentage of participants completing each ABC session, reading the Macmillan booklet (in the control arm), and completing outcome measures at each assessment. This will additionally help calculate the sample size for the proposed follow-on RCT.
* Participants' experience of randomisation to either the intervention or control arm and their experience of being in these arms.
* Participants' responses and feedback to self-complete measures. This will determine suitability of the measures for an RCT.
* Adaptation and testing of a measure of health and social care service use: Assessment of comprehensiveness of the service use measure and acceptability of the measure to collect data for a health economic evaluation

DESIGN

The study will be a parallel, two-arm, RCT, with monitoring of recruitment and retention and an embedded qualitative component to assess feasibility and acceptability of the research process and ABC.

As this is a feasibility study, the objective is not to power the study enough to detect significant differences, but rather, to provide estimates of parameters to inform a subsequent RCT to evaluate intervention effectiveness. Therefore, a formal a-priori power calculation is not needed. The intention is to recruit N = 120 (60 per arm), with participants individually randomised to either the intervention arm (ABC + Macmillan body image booklet) or control arm (Macmillan body image booklet).

RECRUITMENT

The investigators plan to have a phased recruitment, prioritising five geographically diverse NHS Participant Identification Centres (PICs): Bristol, Leeds, Manchester, Nottingham, and Liverpool. To encourage greater diversity of participants, the investigators will additionally advertise the study via various UK cancer support organisations (e.g., Breast Cancer Now, Maggie's). To engage women from underserved groups, the investigators will also advertise the study via OUTpatients (supporting LGBTQIA+ individuals who have had cancer) and the Black Women Rising (supporting women of colour who have had cancer). If these recruitment avenues do not result in obtaining the sample of 120 women, the investigators will use social media as an additional option for recruitment. First, the investigators will advertise the study via the research team's respective university and professional social media channels If this fails to recruit the number of women needed, the last option will involve asking UK-based social media content creators who have had breast cancer (i.e., women from the general public who share their experience of breast cancer with a large group of followers) to advertise the research.

BASELINE DATA COLLECTION

Once participants have provided informed consent, they will complete a series of self-report questionnaires at baseline (i.e., T1, Week 1). These will include demographic and breast cancer-related questions as well as self-report validated measures relating to body image, intimacy, quality of life, functional impairment, and service use. These can be completed either online via Qualtrics or on paper, as per the participant's preference.

RANDOMISATION

After baseline data collection, participants will be randomised to either the intervention or control arm using Sealed Envelope, a web-based randomisation system. Randomisation (at the individual level) will be independent and concealed, using permuted block randomisation. The system will send an email to the Study Manager and CI outlining allocated arms for each participant. The allocation will be made known to the participant via their preferred form of contact (post, email, or telephone).

INTERVENTION AND CONTROL ARM

Irrespective of allocated condition, all participants will be sent Macmillan's freely available psychoeducational body image booklet, which provides support and guidance relating to managing body image concerns. It explains the effects of cancer on body image, and provides practical guidance (e.g., make-up) and psychoeducational guidance (e.g., managing others' reactions), in addition to some CBT strategies.

For intervention arm participants, they will be informed of the next available date to begin ABC. ABC comprises seven 2-hour group sessions (with approximately 8 women per group) delivered online via Microsoft Teams and across 7 consecutive weeks. Rooted in Cognitive Behavioural Therapy, ABC uses strategies to alter unhelpful thoughts, reduce anxiety, and promote non-avoidant behaviours. Other topics are also explored, including sociocultural pressures for women, intimacy, physical activity, self-care, mindfulness, and relaxation. The sessions will be guided using PowerPoint slides, which will include text, images, and videos. Each session will include individual and group-based activities, and participants will be asked to complete between-session readings and activities.

FOLLOW-UP DATA COLLECTION

At T2 (Immediate post-intervention, Week 9), all participants will be asked to complete a series of self-report validated measures relating to body image, intimacy, and quality of life. Participants in the intervention arm will also be asked a series of self-report questions relating to their experience and thoughts on the ABC programme.

At T3 (Three-month post-intervention, Week 20), all participants will be asked to complete a series of self-report validated measures relating to body image, intimacy, quality of life, functional impairment, and service use.

At T4 (Six-month post-intervention, Week 32), all participants will be asked to complete a series of self-report validated measures relating to body image, intimacy, quality of life, functional impairment, and service use. Participants in both arms will also be asked a series of self-report questions relating to their experience of the study and research process (e.g., recruitment, randomisation, the Macmillan body image booklet, communication from the research team throughout the study, and completion of outcome measures).

INTERVIEWS

Purposive sampling will be used to recruit a subset of 16-20 study participants to participate in semi-structured interviews. These interviews will explore the experiences of participants from both conditions in relation to recruitment, randomisation, the Macmillan body image booklet, communication from the research team throughout the study, and completion of outcome measures. Participants from the intervention arm will also be asked about the acceptability of the ABC intervention.

The investigators will target participants at different stages of the study and who may have had different experiences, which will enable us to identify barriers and solutions to participation and retention.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a woman.
* 18+ years old.
* Finished active treatment for breast cancer (including chemotherapy, radiotherapy, targeted and immunotherapy) for breast cancer. There is no time limit on when they finished this treatment. Women on endocrine therapy are eligible to take part. Women with metastatic disease are eligible to take part if on endocrine therapy only.
* Completed primary oncological breast cancer surgery with breast conserving surgery or mastectomy with or without immediate definitive breast reconstruction. Women awaiting delayed breast reconstruction, revision or contralateral symmetrisation surgery are eligible to take part provided this surgery is not planned within the duration of the study.
* Recognises that they are experiencing BID as a result of treatment (regarding how the body looks and/or feels).
* Has the capacity to provide informed consent or supported informed consent (e.g., with a family member/friend).
* Has sufficient understanding of English (as the intervention content and measures are currently only available in English).

Exclusion Criteria:

* Still undergoing active treatment for breast cancer (e.g., oncological breast surgery including those awaiting the second stage of planned expander/implant reconstruction, chemotherapy, targeted therapies, radiotherapy).
* Undergoing exploration for cancer recurrence.
* Has not received a diagnosis of breast cancer e.g., has had prophylactic treatment for a gene mutation (such as risk-reducing mastectomy).
* Has an eating disorder.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self identify as a woman
Enrollment: 120 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Baseline (T1; Week 1)
  The number of women who are recruited into the study, with attention to the method by which women were recruited and their demographic diversity.
Response rates - Self-report outcome measures | Baseline (T1; Week 1), Immediate post-intervention (T2, Week 9), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  The proportion of women who complete the self-report measures at each time point.
Response rates - Intervention arm | Baseline to immediate post-intervention (T1; Week 1 - T2; Week 9)
  the proportion of women completing ABC (the number of sessions attended and the number of between-session activities completed)
Response rates - Control arm | Baseline (T1; Week 1) to 6-month post-intervention (T4; Week 32)
  The proportion of participants in the control arm reading the Macmillan body image booklet (plus the percentage of booklet read)
Quantitative assessment of acceptability - ABC | Immediate post-intervention (T2; Week 9)
  Rating scale relating to the acceptability of the ABC course (e.g., the group format, online nature, between-session activities). Completed by those in intervention arm only.
Quantitative assessment of acceptability - Research process | 6-month post-intervention (T4; Week 32)
  Rating scale to explore acceptability of the research process generally (e.g., information provided about the study, randomisation process, questionnaires) - to be completed by all participants
Qualitative assessment of acceptability - ABC (Open-ended questions) | Immediate post-intervention (T2; Week 9)
  Open-ended questions asking about the acceptability of the ABC course (e.g., the group format, online nature, between-session activities) - to be completed at immediate post-intervention (T2) by participants in the intervention group only.
Qualitative assessment of acceptability - ABC (interviews | Immediate post-intervention (T2; Week 9) to 6-month post-intervention (T4; Week 32)
  Interviews of participant in the intervention group will include questions asking about the acceptability of the ABC course. Interviews will occur across the study period.
Qualitative assessment of acceptability - Research process (Open-ended questions) | 6-month post-intervention (T4; Week 32)
  Open-ended questions to explore acceptability of the research process generally (e.g., information provided about the study, randomisation process, questionnaires) - to be completed by all participants in the six-month post-intervention assessment
Qualitative assessment of acceptability - Research process (interviews) | Baseline (T1; Week 1) to 6-month post-intervention (T4; Week 32)
  All interviews will include questions asking about the acceptability of the research process. Interviews will occur across the study period.
Qualitative assessment of acceptability - ABC course facilitators | Immediate post-intervention (T2; Week 9) to 6-month post-intervention (T4; Week 32)
  All ABC facilitators will also be interviewed following intervention delivery to explore their experience of the programme, as well as their perceived barriers to participant retention, and solutions.

SECONDARY OUTCOMES:
Kessler Psychological Distress Scale (Kessler et al., 2002) | Baseline (T1; Week 1), Immediate post-intervention (T2, Week 9), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  A measure of non-specific psychological distress. Participants are asked to rate their emotional states on a 5-point scale over 10 items. Minimum score is 10, maximum is 50, with higher scores indicating higher levels of psychological distress.
Body Appreciation Scale-2 (Tylka & Wood-Barcalow, 2015) | Baseline (T1; Week 1), Immediate post-intervention (T2, Week 9), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  A measure of a person's acceptance and/or favourable opinions towards their body. Participants are asked to rate each of the 13 items on a 5-point scale. Minimum score is 13, maximum is 65, with higher scores indicating higher levels of body appreciation.
Functional Assessment of Cancer Therapy - Breast (FACT-B Version 4): Breast Cancer Subscale (Brady et al., 1997) | Baseline (T1; Week 1), Immediate post-intervention (T2, Week 9), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  A measure of health-related quality of life for breast cancer patients and includes five subscales. We will be using the Breast Cancer Subscale, whereby participants rate each of the 10 items on a 5-point scale. Minimum score is 0, maximum is 40, with higher scores indicating poorer outcomes.
Hopwood Body Image Scale (Hopwood et al., 2001) | Baseline (T1; Week 1), Immediate post-intervention (T2, Week 9), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  A 10-item scale measuring body image in cancer patients. The scale includes measurement of affective, behavioural, and cognitive elements of body image. Participants rate each item on a 4-point scale. Minimum score is 0, maximum is 30, with higher scores indicating poorer outcomes.
BREAST-Q: Sexual Well-Being Scale (Pusic et al., 2009) | Baseline (T1; Week 1), Immediate post-intervention (T2, Week 9), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  The BREAST-Q is a measure of quality of life and patient satisfaction comprising six subscales, of which we will use only the sexual well-being subscale. This six-item subscale asks participants to rate their feelings related to their sexual attractiveness, sexual confidence, and comfort during sex on a 5 point scale. Minimum score is 6, maximum is 30, with higher scores indicating better outcomes.
Modified version of the Adult Service Use Schedule (AD-SUS; Strauss et al., 2020; Richards et al., 2016). | Baseline (T1; Week 1), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  The AD-SUS is a measure of health and social care service use. Participants indicate which services they have used in the last three months from the list provided (e.g. overnight hospital stay, hospital outpatients appointment, community services). Each of these services has a cost associated with it, and so a cost is calculated for each participant.
  The AD-SUS has been successfully used in depression-focused studies. We have adapted a version of the AD-SUS to ensure coverage of services relevant to women treated for breast cancer. These adaptations where decided through a literature review (existing economic evaluations focused on this population), review of cancer-focused service use measures in the Database of Instruments for Resource Use Measurement (DIRUM; https://www.dirum.org/) and discussions with the team.
Health-related Quality of Life: EQ-5D-5L (Herdman et al., 2011) | Baseline (T1; Week 1), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  A standardised measure of health status, that assesses the respondent's health-related quality of life across five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item is rated between 1 and 5, with higher scores indicating poorer outcomes.
  It also includes a 0-100 visual analogue scale to assess the respondent's overall current health, with higher scores indicating better health.
Recovering Quality of Life-Utility Index (ReQoL-10; Keetharuth et al., 2018) | Baseline (T1; Week 1), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  Measure of psychological wellbeing where participants are asked to rate their thoughts, feelings and activities over the last week. For each statement they are asked to select from the following five options: None of the time, Only occasionally, Sometimes, Often, Most or all of the time.
  Minimum score is 0, maximum is 44, with higher scores indicating better outcomes.
Work and Social Adjustment Scale (WSAS; Mundt et al., 2002) | Baseline (T1; Week 1), 3-month post-intervention (T3; Week 20), 6-month post-intervention (T4; Week 32)
  Assesses the impact of a person's psychological wellbeing on their ability to function in terms of work, home management, social leisure, private leisure and personal or family relationships. There are 5 items which participants are asked to rate on a 9-point scale. Minimum score is 0, maximum is 40, with higher scores indicating poorer outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Lewis-Smith, Principal Investigator — University of the West of England
Locations (1):
- Centre for Appearance Research, University of the West of England, Bristol, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
When publishing the findings of the research, a data sharing statement will be shared, which will state that researchers can contact the research team to enquire about accessing the underpinning research data. Data access requests will be managed following UWE Bristol policies and practices, and release of data will be subject to a data use agreement between UWE Bristol and the third party requesting the data.

REFERENCES:
- [Background] Begovic-Juhant A, Chmielewski A, Iwuagwu S, Chapman LA. Impact of body image on depression and quality of life among women with breast cancer. J Psychosoc Oncol. 2012;30(4):446-60. doi: 10.1080/07347332.2012.684856. PMID 22747107
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3(2), 77-101. https://doi.org/10.1191/1478088706qp063oa
- [Background] Braun, V. and Clarke, V. (2022) Conceptual and design thinking for thematic analysis. Qualitative Psychology. 9(1): p. 3.
- [Background] Carreira H, Williams R, Funston G, Stanway S, Bhaskaran K. Associations between breast cancer survivorship and adverse mental health outcomes: A matched population-based cohort study in the United Kingdom. PLoS Med. 2021 Jan 7;18(1):e1003504. doi: 10.1371/journal.pmed.1003504. eCollection 2021 Jan. PMID 33411711
- [Background] Cash, T.F. and Pruzinsky, T. (2002). Body image: a handbook of theory, research, and clinical practice. New York: Guilford Publications.
- [Background] Cohen M, Anderson RC, Jensik K, Xiang Q, Pruszynski J, Walker AP. Communication between breast cancer patients and their physicians about breast-related body image issues. Plast Surg Nurs. 2012 Jul-Aug;32(3):101-5. doi: 10.1097/PSN.0b013e3182650994. PMID 22929196
- [Background] Cousson-Gelie F, Bruchon-Schweitzer M, Dilhuydy JM, Jutand MA. Do anxiety, body image, social support and coping strategies predict survival in breast cancer? A ten-year follow-up study. Psychosomatics. 2007 May-Jun;48(3):211-6. doi: 10.1176/appi.psy.48.3.211. PMID 17478589
- [Background] Davis C, Tami P, Ramsay D, Melanson L, MacLean L, Nersesian S, Ramjeesingh R. Body image in older breast cancer survivors: A systematic review. Psychooncology. 2020 May;29(5):823-832. doi: 10.1002/pon.5359. Epub 2020 Feb 20. PMID 32048373
- [Background] Falk Dahl CA, Reinertsen KV, Nesvold IL, Fossa SD, Dahl AA. A study of body image in long-term breast cancer survivors. Cancer. 2010 Aug 1;116(15):3549-57. doi: 10.1002/cncr.25251. PMID 20564138
- [Background] Helms RL, O'Hea EL, Corso M. Body image issues in women with breast cancer. Psychol Health Med. 2008 May;13(3):313-25. doi: 10.1080/13548500701405509. PMID 18569899
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Hopwood P, Fletcher I, Lee A, Al Ghazal S. A body image scale for use with cancer patients. Eur J Cancer. 2001 Jan;37(2):189-97. doi: 10.1016/s0959-8049(00)00353-1. PMID 11166145
- [Background] Keetharuth AD, Brazier J, Connell J, Bjorner JB, Carlton J, Taylor Buck E, Ricketts T, McKendrick K, Browne J, Croudace T, Barkham M. Recovering Quality of Life (ReQoL): a new generic self-reported outcome measure for use with people experiencing mental health difficulties. Br J Psychiatry. 2018 Jan;212(1):42-49. doi: 10.1192/bjp.2017.10. PMID 29433611
- [Background] Keetharuth AD, Rowen D, Bjorner JB, Brazier J. Estimating a Preference-Based Index for Mental Health From the Recovering Quality of Life Measure: Valuation of Recovering Quality of Life Utility Index. Value Health. 2021 Feb;24(2):281-290. doi: 10.1016/j.jval.2020.10.012. Epub 2020 Nov 27. PMID 33518035
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Lam WW, Li WW, Bonanno GA, Mancini AD, Chan M, Or A, Fielding R. Trajectories of body image and sexuality during the first year following diagnosis of breast cancer and their relationship to 6 years psychosocial outcomes. Breast Cancer Res Treat. 2012 Feb;131(3):957-67. doi: 10.1007/s10549-011-1798-2. Epub 2011 Oct 5. PMID 21971728
- [Background] Lewis-Smith, H. (2017). Body image in midlife: Developing a psychosocial intervention for women who have received treatment for breast cancer. University of the West of England.
- [Background] Lewis-Smith H, Diedrichs PC, Harcourt D. A pilot study of a body image intervention for breast cancer survivors. Body Image. 2018 Dec;27:21-31. doi: 10.1016/j.bodyim.2018.08.006. Epub 2018 Aug 16. PMID 30121489
- [Background] Lewis-Smith H, Diedrichs PC, Rumsey N, Harcourt D. A systematic review of interventions on body image and disordered eating outcomes among women in midlife. Int J Eat Disord. 2016 Jan;49(1):5-18. doi: 10.1002/eat.22480. Epub 2015 Nov 26. PMID 26607999
- [Background] Lewis-Smith H, Diedrichs PC, Rumsey N, Harcourt D. Efficacy of psychosocial and physical activity-based interventions to improve body image among women treated for breast cancer: A systematic review. Psychooncology. 2018 Dec;27(12):2687-2699. doi: 10.1002/pon.4870. Epub 2018 Oct 2. PMID 30161285
- [Background] Lewis-Smith H, Diedrichs PC, Bond R, Harcourt D. Psychological and sociocultural influences on body image among midlife women with and without a history of breast cancer: Testing the Tripartite Influence Model of Body Image. Body Image. 2020 Dec;35:114-125. doi: 10.1016/j.bodyim.2020.08.011. Epub 2020 Sep 30. PMID 33010788
- [Background] Mausbach BT, Decastro G, Schwab RB, Tiamson-Kassab M, Irwin SA. Healthcare use and costs in adult cancer patients with anxiety and depression. Depress Anxiety. 2020 Sep;37(9):908-915. doi: 10.1002/da.23059. Epub 2020 Jun 2. PMID 32485033
- [Background] McWilliam CL, Brown JB, Stewart M. Breast cancer patients' experiences of patient-doctor communication: a working relationship. Patient Educ Couns. 2000 Feb;39(2-3):191-204. doi: 10.1016/s0738-3991(99)00040-3. PMID 11040719
- [Background] Moreira H, Canavarro MC. A longitudinal study about the body image and psychosocial adjustment of breast cancer patients during the course of the disease. Eur J Oncol Nurs. 2010 Sep;14(4):263-70. doi: 10.1016/j.ejon.2010.04.001. Epub 2010 May 21. PMID 20493769
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] O'Cathain A, Hoddinott P, Lewin S, Thomas KJ, Young B, Adamson J, Jansen YJ, Mills N, Moore G, Donovan JL. Maximising the impact of qualitative research in feasibility studies for randomised controlled trials: guidance for researchers. Pilot Feasibility Stud. 2015 Sep 7;1:32. doi: 10.1186/s40814-015-0026-y. eCollection 2015. PMID 27965810
- [Background] Paterson CL, Lengacher CA, Donovan KA, Kip KE, Tofthagen CS. Body Image in Younger Breast Cancer Survivors: A Systematic Review. Cancer Nurs. 2016 Jan-Feb;39(1):E39-58. doi: 10.1097/NCC.0000000000000251. PMID 25881807
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Richards DA, Ekers D, McMillan D, Taylor RS, Byford S, Warren FC, Barrett B, Farrand PA, Gilbody S, Kuyken W, O'Mahen H, Watkins ER, Wright KA, Hollon SD, Reed N, Rhodes S, Fletcher E, Finning K. Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): a randomised, controlled, non-inferiority trial. Lancet. 2016 Aug 27;388(10047):871-80. doi: 10.1016/S0140-6736(16)31140-0. Epub 2016 Jul 23. PMID 27461440
- [Background] Rosman S. Cancer and stigma: experience of patients with chemotherapy-induced alopecia. Patient Educ Couns. 2004 Mar;52(3):333-9. doi: 10.1016/S0738-3991(03)00040-5. PMID 14998604
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Strauss C, Arbon A, Barkham M, Byford S, Crane R, de Visser R, Heslin M, Jones AM, Jones F, Lea L, Parry G, Rosten C, Cavanagh K. Low-Intensity Guided Help Through Mindfulness (LIGHTMIND): study protocol for a randomised controlled trial comparing supported mindfulness-based cognitive therapy self-help to supported cognitive behavioural therapy self-help for adults experiencing depression. Trials. 2020 May 4;21(1):374. doi: 10.1186/s13063-020-04322-1. PMID 32366320
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Van Beek FE, Wijnhoven LMA, Holtmaat K, Custers JAE, Prins JB, Verdonck-de Leeuw IM, Jansen F. Psychological problems among cancer patients in relation to healthcare and societal costs: A systematic review. Psychooncology. 2021 Nov;30(11):1801-1835. doi: 10.1002/pon.5753. Epub 2021 Jul 6. PMID 34228838
- [Derived] Lewis-Smith H, Jones A, White P, Byford S, Fairbrother P, Potter S, Harcourt D. Accepting your Body after Cancer (ABC), a group-based online intervention for women treated for breast cancer: study protocol for a feasibility randomised controlled trial. BMJ Open. 2025 Jan 22;15(1):e097817. doi: 10.1136/bmjopen-2024-097817. PMID 39843373